# Statistical Analysis Plan for the study: "Effects of menaquinone-7 supplementation in patients with aortic valve calcification"

SAP authors: Axel Diederichsen<sup>a</sup>, Selma Hasific<sup>a</sup>, Lars Folkestad<sup>b</sup>, Jes Lindholt<sup>c</sup>, Jordi Dahl<sup>a</sup>, Kristian Øvrehus<sup>a</sup>, Sören Möller<sup>d</sup>

#### Affiliations:

Primary publication: Change in AVC score

Secondary publication: Change in aortic calcification and diameter

P13

Secondary publication: Change in coronary artery calcification and plaque composition

P19

Secondary publication: Changes in volumetric bone mineral density

P31

### Introduction

This document specifies the planned statistical analysis for the study "Effects of menaquinone-7 supplementation in patients with aortic valve calcification: study protocol for a randomised controlled trial" as carried out following the protocol published in BMJ Open (1).

### Sample size considerations

According to the protocol (1): "The study was designed to have 80% power to detect a 20 % difference in progression of aortic valve calcification score between the treatment groups. At least 354 patients were required for the study to be conclusive, and we planned to include 400 patients."

### Randomizations

Subjects were be randomized 1:1 stratified by site (Odense University Hospital - Odense, Svendborg Hospital, Vejle Hospital or Silkeborg Hospital) and AVC score (300–599 or ≥600).

<sup>&</sup>lt;sup>a</sup> Department of Cardiology, Odense University Hospital, Odense, Denmark

<sup>&</sup>lt;sup>c</sup> Department of Endocrinology, Odense University Hospital, Odense, Denmark

<sup>&</sup>lt;sup>c</sup> Department of Cardiothoracic and Vascular Surgery, Odense University Hospital, Odense, Denmark

<sup>&</sup>lt;sup>d</sup> OPEN – Open Patient data Explorative Network, Odense University Hospital and Department of Clinical Research, University of Southern Denmark, Odense, Denmark

### Interim analyses

During conduct of the study, an interim analysis was conducted to determine if the intervention should be prolonged by 6 months. The interim analyses concluded that this was not necessary. As the interim analysis did only influence how the intervention was performed, but neither sample size nor possible discontinuation of the study, we did not take the interim analysis into account in the final analyses.

### Statistical principles

All analyses were performed in the intention-to-treat population and as superiority analyses. Two-sided p-values of 0.05 or less were considered to indicate statistical significance and associations and effect estimates will be reported with 95% probability symmetric confidence interval (2.5% to 97.5% quantile).

### Practical considerations

Data were collected using REDCap (2, 3) hosted by OPEN (Open Patient data Explorative Network, Odense University Hospital, Odense Denmark) with project number OP\_530. Data were analyzed using Stata (4) on OPEN's secure analysis server (OPEN Analyse). A prespecified random seed of 7042021 will be used for bootstrapping and imputation.

### Planned analyses for primary publication: Change in AVC score

### Exclusion criteria

Participants with AVC < 300 at baseline will be excluded from all analyses in this publication.

### Outcomes

### Primary outcome: Main analysis

The primary outcome was the change in aortic valve calcification (AVC) score (numerical) from baseline to 24 month for the full cohort of included patients.

### Secondary outcomes to be included in the primary publication

### Secondary outcomes were

- Change in AVC from baseline to 24 months in two prespecified subgroups (baseline AVC score 300-599 and ≥600).
- Change in AVC from baseline to 12 months and from 12 months to 24 months, both for the full cohort as well as for the two subgroups.
- Changes in aortic valve area from baseline to 24 months (numerical)
- Change in peak aortic-jet velocity from baseline to 24 months (numerical)
- Need of heart valve surgery (dichotomous, occurred / not occurred between baseline and 24 months)

- Change in MGP with different phosphorylation and carboxylation forms (numerical)
- Change in QoL from baseline to 24 months (numerical)

### Safety outcomes

### Safety outcomes were

- Death (all cause and cardivascular cause) (dichotomous)
- Cardiovascular events (a composite endpoint of myocardial infarction, coronary revascularization, stroke, aortic disease, significant peripheral artery disease (surgery), as well as these endpoints separately) (all dichotomous)
- Progressive aortic valve disease (more than 50% increase in AVC score) (dichotomous)
- Venous thromboembolism (dichotomous)
- Severe bleeding
- Low energy or spontaneous fracture
- Cancer (recurrent cancer or new cancer) (dichotomous)
- The following laboratory measurements: hemoglobin, leucocytes, thrombocytes, albumin, creatinine (eGFR), urea, calcium, phosphate, magnesium, troponine, creatine kinase, alanine aminotransferase, lactate dehydrogenase, bilirubin, alkaline phosphatase, total-cholesterol, low-density lipoprotein, high-density lipoprotein, parathyroid hormone, vitamin D, prothrombin time-international normalised ratio (PT-INR) and activated partial thromboplastin time (all numerical)

Dichotomous safety outcomes were evaluated as occurred / not occurred between baseline and 24 months. Numerical safety outcomes were evaluated as change from baseline to 12 and 24 months.

### Planned tables and figures and corresponding analyses

### Table 1. Characteristics of patients at baseline

Characteristics (as listed in Table 1 below, numerical characteristics marked with [numerical]) of patients at baseline will be reported separately for the two treatment groups. Characteristics will be reported as

- Mean and standard deviation (SD) for numerical characteristics, which are approximately
  normally distributed in both treatment groups as investigated by normal quantile-quantile
  plots. These characteristics will be compared between groups by two-sample t-test with
  assumed equal variance, or with assumed unequal variance if indicated by Levene's test for
  equality of variance (5).
- Median and 1<sup>st</sup> and 3<sup>rd</sup> quartile (inter quartile range (IQR)) for numerical characteristics, which
  are not approximately normally distributed in at least one treatment group as indicated by
  normal quantile-quantile plots. These characteristics will be compared between groups by
  Wilcoxon rank-sum test.

• Counts and proportions for categorical characteristics (with categories as specified in Table 1 below). These characteristics will be compared between groups by  $\chi^2$ -test if all counts are at least 5, or with Fisher's exact test otherwise.

No adjustments for multiple testing will be carried out in Table 1 and no effect sizes for differences between groups will be estimated. Missing observations will be excluded from tests in Table 1, and number of missing observations in each group will be specified.

| Characteristic | Vitamin K +D group<br>(N=XX) | Placebo group<br>(N=XX) | P-value |
|---|---|---|---|
| Age – years [numerical] | , , | , , | |
| Baseline AVC – AU [numerical] | | | |
| Echocardiography | | | |
| Bicuspid aortic valve – no (%) | | | |
| V <sub>max</sub> - cm/sec [numerical] | | | |
| Aortic valve area - cm² [numerical] | | | |
| • Left ventricular ejection fraction -% [numerical] | | | |
| Estimated GFR – ml/min/1.73 m² [numerical] | | | |
| dp-ucMGP – pmol/L [numerical] | | | |
| Body-mass index [numerical] | | | |
| Systolic Blood pressure – mmHg [numerical] | | | |
| Smoking | | | |
| Active smokers - no (%) | | | |
| Former smokers – no (%) | | | |
| Non-smokers – no (%) | | | |
| Coexisting condition – no (%) | | | |
| Hypertension | | | |
| Diabetes | | | |
| Ischemic heart disease | | | |
| Atrial fibrillation | | | |
| Renal failure (eGFR<60) | | | |
| Medications – no (%) | | | |
| ACE inhibitor or ARB | | | |
| Beta-blocker | | | |
| Mineralocorticoid-receptor antagonist | | | |
| Antiplatelet therapy | | | |
| NOAC | | | |
| Statin therapy ACT to the state of the | | diam da maMCD danha | |

ACE denotes angiotensin-converting enzyme, ARB angiotensin-receptor blocker, AVC aortic valve calcification, dp-ucMGP dephosphorylated-uncarboxylated Matrix Gla-Protein, GFR glomerular filtration rate, NOAC new-onset anticoagulant † The body-mass index is the weight in kilograms divided by the square of the height in meters.

### Table 2. Primary outcome and numerical secondary outcomes

Primary outcome and numerical secondary outcomes will be analyzed by mixed effects linear regression. The mixed effects linear regression models will include a fixed effect for treatment, a fixed effect for time point (baseline, 12 and 24 months) and a fixed effects interaction between treatment and time point. As baseline measurements are obtained before randomization, treatment at baseline will be modelled as a

separate common treatment category, constraining baseline measurements to no systematic treatment effect between the two treatment arms, as suggested in literature (6). All mixed effects models will include a random intercept for each included patient. Normality assumptions on residuals and random effects will be evaluated by normal quantile-quantile plots. In case deviations from normality assumptions are detected analyses will be repeated with nonparametric bootstrapping with 1,000 bootstrapping samples (handling individual patients as bootstrapping clusters, and treatment groups as bootstrapping strata).

Missing data will be excluded from analyses in Table 2 (but see sensitivity analyses below).

| | | Vitamin K +D<br>group | Placebo group | | |
|---|---|---|---|---|---|
| | | Mean change<br>from baseline (95<br>% CI) | Mean change<br>from baseline<br>(95 % CI) | Treatment effect<br>(95 % CI) | P-value |
| Primary outcome: Ma | ain analysis | , | , | | |
| AVC score (all patients) | 0 – 24 months | | | | |
| Numerical secondary | outcomes | 1 | | | 1 |
| AVC score (all | 0 – 12 months | | | | |
| patients) | 12 – 24 | | | | |
| | months | | | | |
| AVC score | 0 – 24 months | | | | |
| (baseline AVC score | 0 – 12 months | | | | |
| 300-599) | 12 – 24 | | | | |
| | months | | | | |
| AVC score | 0 – 24 months | | | | |
| (baseline AVC score | 0 – 12 months | | | | |
| ≥600) | 12 – 24 | | | | |
| | months | | | | |
| Aortic valve area | 0 – 24 months | | | | |
| Peak aortic-jet | 0 – 24 months | | | | |
| velocity | | | | | |
| dp-ucMGP | 0 – 24 months | | | | |
| QoL | 0 – 24 months | | | | |

Table 3. Dichotomous secondary outcomes and adverse events

Dichotomous secondary outcomes (valvular surgery between baseline and 24 months) and adverse events are reported as counts and proportions separately for each treatment group and compared between groups by  $\chi^2$ -test if all counts are at least 5, or with Fisher's exact test otherwise. If a patient reported multiple events of the same outcomes, this will be handled dichotomously as experiencing the outcome in the analyses, but the count of such patients will be reported in a parenthesis or footnote to the table.

Missing observations will be excluded from tests in Table 2, and number of missing observations in each group will be specified.

| Event | Vitamin K +D group | Placebo group | p-value |
|-------|--------------------|---------------|---------|
|-------|--------------------|---------------|---------|

| | (N=XX) | (N=XX) |
|-------------------------------------------------|--------|--------|
| Outcome | | |
| Valvular Surgery – no (%) | | |
| Adverse Events | | |
| Any event – no (%) | | |
| Death – no (%) | | |
| Cardiovascular events (combined) – no (%) | | |
| Myocardial infarction | | |
| Coronary revascularization | | |
| Stroke | | |
| Aortic disease | | |
| Peripheral artery surgery | | |
| Progressive aortic valve disease (more than 50% | | |
| increase in AVC score) | | |
| Severe bleeding – no (%) | | |
| Venous thromboembolism – no (%) | | |
| Low energy fracture– no (%) | | |
| Incident cancer – no (%) | | |

### Table 4. Numerical safety outcomes

Numerical safety outcomes will be analyzed by linear mixed models corresponding to the analyses specified for the primary outcome in Table 2. No subgroup analyses will be performed.

| | | Vitamin K +D group | Placebo group | | |
|---|---|---|---|---|---|
| | | Mean change (95 % | Mean change | Treatment | P- |
| | | CI) | (95 % CI) | effect (95 % CI) | value |
| hemoglobin | 0 - 24 months | | | | |
| creatinine (eGFR) | 0 - 24 months | | | | |
| calcium | 0 - 24 months | | | | |
| phosphate | 0 - 24 months | | | | |
| parathyroid hormone | 0 - 24 months | | | | |
| vitamin D | 0 - 24 months | | | | |
| activated partial | 0 - 24 months | | | | |
| thromboplastin time | | | | | |
| prothrombin time- | 0 - 24 months | | | | |
| international | | | | | |
| normalised ratio (PT- | | | | | |
| INR) | | | | | |

### Table 5. Stratified analyses of the primary outcome

Analyses of the primary outcome (AVC score) will be repeated stratifying for age (<70 or ≥70 years at baseline), diabetes (yes / no at baseline), hypertension (yes / no at baseline), atrial fibrillation (yes / no at baseline), ischemic heart disease (yes / no at baseline), renal failure (yes / no at baseline), statin therapy (yes / no at baseline), and MGP (below / above median). In these analyses, patients will not be stratified by baseline AVC score 300-599 and ≥600. The same models as for Table 2 will be applied for these analyses.

| | Vitamin K +D group | Placebo group | | |
|---|---|---|---|---|
| | Mean change from baseline (95 % CI) | Mean change<br>from baseline<br>(95 % CI) | Treatment effect<br>(95 % CI) | P-value |
| Age < 70 years | | | | |
| Age ≥70 years | | | | |
| No diabetes | | | | |
| Diabetes | | | | |
| No | | | | |
| hypertension | | | | |
| Hypertension | | | | |
| No atrial | | | | |
| fibrillation | | | | |
| Atrial | | | | |
| fibrillation | | | | |
| No ischemic | | | | |
| heart disease | | | | |
| Ischemic heart | | | | |
| disease | | | | |
| No renal failure | | | | |
| Renal failure | | | | |
| No statin | | | | |
| therapy | | | | |
| Statin therapy | | | | |
| Baseline MGP < | | | | |
| median | | | | |
| Baseline MGP | | | | |
| >= median | | | | |

### Supplementary Table S1. Sensitivity analysis: Primary outcome and numerical secondary outcomes with imputation

If more than 5% of observations are missing at 24 months for the main analysis of the primary outcome reported in Table 2 the analysis will be repeated using multiple imputation (assuming missing at random) by linear regression with all baseline characteristics included in Table 1 as covariates generating 100 imputation. Results will be reported in a table structured as Table 2.

### Supplementary Table S2. Sensitivity analysis: Primary outcome on subgroup with high compliance

The analysis of primary outcome (all patients 0-24 months) will be repeated (with the same methodology as specified for Table 3) on those patients, who reported a compliance of at least 90% during the study period. Furthermore, number and proportion of patients included in this analysis will be reported in Table S4, together with odds ratio (with 95% confidence interval) and p-value determined by univariate logistic regression for difference in compliance rate between treatment arms will be reported.

| | | Vitamin K +D group | Placebo group | Group difference | |
|---|---|---|---|---|---|
| | | Number (proportion) | Number<br>(proportion) | Odds ratio (95 % CI) | P-value |
| Compliance of a | ıl<br>at least 90% | (ριοροιτίση) | (proportion) | Cij | |
| | | Mean change from baseline (95 % CI) | Mean change<br>from baseline<br>(95 % CI) | Treatment effect<br>(95 % CI) | P-value |
| Primary outcom | Primary outcome (only including with compliance of at least 90%) | | | | |
| AVC score (all patients) | 0 – 24 months | | | | |

### Supplementary Table S3. Safety outcomes of clinical biochemistry

Numerical safety outcomes will be analyzed by linear mixed models corresponding to the analyses specified for the primary outcome in Table 2. No subgroup analyses will be performed.

| | | Vitamin K +D | Placebo | | |
|---|---|---|---|---|---|
| | | group | group | | |
| | | Mean change (95 | Mean change | Treatment | P-value |
| | | % CI) | (95 % CI) | effect (95 % CI) | |
| hemoglobin | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| leucocytes | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| thrombocytes | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| albumin | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| creatinine (eGFR) | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| urea | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| calcium | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| magnesium | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| phosphate | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| troponine | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| creatine kinase | 0 - 12 months | | | | |
| | 0 - 24 months | | | | |
| alanine | 0 - 12 months | | | | |
| aminotransferase | 0 - 24 months | | | | |
| lactate | 0 - 12 months | | | | |
| dehydrogenase | 0 - 24 months | | | | |
| bilirubin | 0 - 12 months | | | | |

| | 0 04 11 |
|-------------------|---------------|
| | 0 - 24 months |
| alkaline | 0 - 12 months |
| phosphatase | 0 - 24 months |
| total-cholesterol | 0 - 12 months |
| | 0 - 24 months |
| low-density | 0 - 12 months |
| lipoprotein | 0 - 24 months |
| high-density | 0 - 12 months |
| lipoprotein | 0 - 24 months |
| triglyceride | 0 - 12 months |
| | 0 - 24 months |
| parathyroid | 0 - 12 months |
| hormone | 0 - 24 months |
| vitamin D | 0 - 12 months |
| | 0 - 24 months |
| prothrombin | 0 - 12 months |
| time- | 0 - 24 months |
| international | |
| normalised ratio | |
| (PT-INR) | |
| activated partial | 0 - 12 months |
| thromboplastin | 0 - 24 months |
| time | |

Figure 1. Enrollment and Randomization of Patients.

Flow chart



### Figure 2. AVC progression according to treatment allocation.

AVC score at baseline, 12, and, 24 months will be presented at line graph for the two treatment groups presenting mean with 95% confidence interval (as obtained from the linear mixed models applied for Table 3). The figure will be presented for all patients (Figure 2A) as well as stratified by the baseline AVC score subgroups 300-599 (Figure 2B) and ≥600 (Figure 2C). (See mockup figure 2A below, 2B and 2C are similar)



Figure 3. AVA (A) and Vmax (B) changes according to treatment allocation

AVA (Figure 3A) and Vmax (Figure 3B) at baseline, 12, and, 24 months will be presented at line graph for the two treatment groups presenting mean with 95% confidence interval (as obtained from the linear mixed models applied for Table 3). (See mockup figures below)



Figure 4. Forest plot of stratified analyses of the primary outcome

Coefficients with 95% confidence intervals from stratified analyses (as reported in Table 4) for differences in primary outcome (change of AVA score from baseline to 24 months) between treatment groups will be presented as a forest plot. (See mockup figure below.)



## Planned analyses for secondary publication: Change in aortic calcification and diameter

### Exclusion criteria

Participants with prior aortic surgery are excluded from this study.

### Outcomes

### Primary outcome

- Co-primary outcome 1: change in aortic calcification score (numerical) from baseline to 24 month.
- Co-primary outcome 2: change in aortic dilatation (numerical) from baseline to 24 month.

### Secondary outcomes

- Change in aortic calcification score from baseline to 12 months and from 12 months to 24 months.
- Change in aortic diameter from baseline to 12 months and from 12 months to 24 months.
- Need of aortic surgery (dichotomous, occurred / not occurred between baseline and 24 months).

### Planned tables and figures and corresponding analyses

### Table 1. Characteristics of patients at baseline

Statistical methods applied for table 1 are similar to the statistics used for table 1 in the primary publication.

| Characteristic | Vitamin K +D group<br>(N=XX) | Placebo group<br>(N=XX) | P-value |
|---|---|---|---|
| Age – years [numerical] | | | |
| Baseline aortic calcification score – AU | | | |
| [numerical] | | | |
| Ascending | | | |
| • Arcus | | | |
| Descending | | | |
| Suprarenal | | | |
| Infrarenal | | | |
| Renal artery | | | |
| Iliaca com artery | | | |
| Iliaca ext artery | | | |
| Baseline aortic diameter – mm [numerical] | | | |
| Ascending | | | |
| • Arcus | | | |
| Descending | | | |
| Infrarenal | | | |
| Estimated GFR – ml/min/1.73 m <sup>2</sup> [numerical] | | | · |
| Body-mass index [numerical] | | | |

| dp-ucMGP – pmol/L |
|--------------------------------------------|
| Systolic Blood pressure – mmHg [numerical] |
| Smoking |
| Active smokers - no (%) |
| Former smokers – no (%) |
| Non-smokers – no (%) |
| Coexisting condition – no (%) |
| Hypertension |
| Diabetes |
| Ischemic heart disease |
| Atrial fibrillation |
| Renal failure (eGFR<60) |
| Medications – no (%) |
| ACE inhibitor or ARB |
| Beta-blocker |
| Mineralocorticoid-receptor antagonist |
| Antiplatelet therapy |
| NOAC |
| Statin therapy |

ACE denotes angiotensin-converting enzyme, ARB angiotensin-receptor blocker, AVC aortic valve calcification, dp-ucMGP dephosphorylated-uncarboxylated Matrix Gla-Protein, GFR glomerular filtration rate, NOAC new-onset anticoagulant † The body-mass index is the weight in kilograms divided by the square of the height in meters.

### Table 2. Primary outcome and numerical secondary outcomes

Primary outcome and numerical secondary outcomes will be analyzed by mixed effects linear regression. The mixed effects linear regression models will include a fixed effect for treatment, a fixed effect for time point (baseline, 12 and 24 months) and a fixed effects interaction between treatment and time point. As baseline measurements are obtained before randomization, treatment at baseline will be modelled as a separate common treatment category, constraining baseline measurements to no systematic treatment effect between the two treatment arms, as suggested in literature (6). All mixed effects models will include a random intercept for each included patient. Normality assumptions on residuals and random effects will be evaluated by normal quantile-quantile plots. In case deviations from normality assumptions are detected analyses will be repeated with nonparametric bootstrapping with 1,000 bootstrapping samples (handling individual patients as bootstrapping clusters, and treatment groups as bootstrapping strata).

Due to the 12 primary outcome measures, we will apply the Bonferroni-Holm-method to adjust for multiple testing of these 12 p-values. The unadjusted p-values will be reported in the table, but it will be indicated by a \* if treatment effects are still significant at the 5% level after Bonferroni-Holm-adjustment. No adjustment for multiple testing will be performed for secondary outcomes.

Missing data will be excluded from analyses in Table 2 (but see sensitivity analyses below).

| | Vitamin K +D | Placebo | | |
|-----------------|--------------|-------------|------------------|---------|
| | group | group | | |
| | Mean change | Mean change | Treatment effect | P-value |
| | (95 % CI) | (95 % CI) | (95 % CI) | |
| Primary outcome | | | | |

| Aortic calcification | 0 – 24 months |
|---|---|
| | 0 – 24 months |
| score | |
| Ascending | |
| • Arcus | |
| Descending | |
| <ul> <li>Suprarenal</li> </ul> | |
| <ul> <li>Infrarenal</li> </ul> | |
| <ul> <li>Renal artery</li> </ul> | |
| <ul> <li>Iliaca com artery</li> </ul> | |
| Iliaca ext artery | |
| Aortic diameter | 0 – 24 months |
| <ul> <li>Ascending</li> </ul> | |
| <ul> <li>Arcus</li> </ul> | |
| <ul> <li>Descending</li> </ul> | |
| <ul> <li>Infrarenal</li> </ul> | |
| Numerical secondary | Numerical secondary outcomes |
| Aortic calcification | 0 – 12 months |
| score | and |
| <ul> <li>Ascending</li> </ul> | 12 – 24 months |
| <ul> <li>Arcus</li> </ul> | |
| <ul> <li>Descending</li> </ul> | |
| <ul> <li>Suprarenal</li> </ul> | |
| <ul> <li>Infrarenal</li> </ul> | |
| Renal artery | |
| Iliaca com artery | |
| Iliaca ext artery | |
| Aortic diameter | 0 – 12 months |
| <ul> <li>Ascending</li> </ul> | and |
| Arcus | 12 – 24 months |
| <ul> <li>Descending</li> </ul> | |
| Infrarenal | |

### Table 3. Dichotomous secondary outcomes

Dichotomous secondary outcome (aortic surgery between baseline and 24 months) is reported as counts and proportions separately for each treatment group and compared between groups by  $\chi^2$ -test if all counts are at least 5, or with Fisher's exact test otherwise. If a patient reported multiple events of the same outcomes, this will be handled dichotomously as experiencing the outcome in the analyses, but the count of such patients will be reported in a parenthesis or footnote to the table.

Missing observations will be excluded from tests in Table 3, and number of missing observations in each group will be specified.

| Event | Vitamin K +D group<br>(N=XX) | Placebo group<br>(N=XX) | p-value |
|---|---|---|---|
| Outcome | | | |
| Aortic surgery – no (%) | | | |

### Table 4. Stratified analyses of the primary outcome

Analyses of the primary outcome (change in aortic calcification score and change in aortic dilatation) will be repeated stratifying for and MGP (below / above median). The same models as for Table 2 will be applied for these analyses.

### Supplementary Table S1. Sensitivity analysis: Primary outcome with imputation

If more than 5% of observations are missing at 24 months for the main analysis of the primary outcome reported in Table 2 the analysis will be repeated using multiple imputation (assuming missing at random) by linear regression with all baseline characteristics included in Table 1 as covariates generating 100 imputation sets. Results will be reported in a table structured as Table 2.

### Supplementary Table S2. Sensitivity analysis: Primary outcome on subgroup with high compliance

The analysis of primary outcome will be repeated (with the same methodology as specified for Table 2) on those patients, who reported a compliance of at least 90% during the study period. Furthermore, number and proportion of patients included in this analysis will be reported in Table S5, together with odds ratio (with 95% confidence interval) and p-value determined by univariate logistic regression for difference in compliance rate between treatment arms will be reported.

| | | Vitamin K +D | Placebo group | Group difference | |
|---|---|---|---|---|---|
| | | group | | | |
| | | | | | T |
| | | Number | Number | Odds ratio (95 | P- |
| | | (proportion) | (proportion) | % CI) | value |
| Compliance of at least 9 | 0% | | | | |
| | | Mean change | Mean change | Treatment | P- |
| | | from baseline | from baseline (95 | effect (95 % CI) | value |
| | | (95 % CI) | % CI) | | |
| Primary outcome (only i | ncluding with co | mpliance of at least | 90%) | | |
| Aortic calcification | 0 – 24 | | | | |
| score | months | | | | |
| <ul> <li>Ascending</li> </ul> | | | | | |
| • Arcus | | | | | |
| <ul> <li>Descending</li> </ul> | | | | | |
| <ul> <li>Suprarenal</li> </ul> | | | | | |
| <ul> <li>Infrarenal</li> </ul> | | | | | |
| Renal artery | | | | | |
| Iliaca com artery | | | | | |
| Iliaca ext artery | | | | | |
| Aortic diameter | 0 – 24 | | | | |
| Ascending | months | | | | |
| • Arcus | | | | | |
| Descending | | | | | |
| Infrarenal | | | | | |

Figure 1. Enrollment and Randomization of Patients.

Flow chart



### Figure 2A-H. Aortic calcification according to treatment allocation.

Aortic calcification score at baseline, 12, and, 24 months will be presented at line graph for the two treatment groups presenting mean with 95% confidence interval (as obtained from the linear mixed models applied for Table 2) for each of the 8 aortic calcification outcomes as Figures 2A to 2I. (See mockup figure 2A below, 2B-I similar)



Figure 3A-D. Aortic diameter according to treatment allocation.

Aortic diameter at baseline, 12, and, 24 months will be presented at line graph for the two treatment groups presenting mean with 95% confidence interval (as obtained from the linear mixed models applied for Table 2) for each of the 4 aortic diameter outcomes as Figures 3A to 3D. (See mockup figure 3A below, 3B-D similar)



# Planned analyses for secondary publication: Change in coronary artery calcification and plaque composition

#### Exclusion criteria

Participants with known cardiovascular disease (CVD) defined as previous acute myocardial infarction (AMI), percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG) surgery will be excluded.

#### Outcomes

### Primary outcome

The primary outcome in this substudy is the change in coronary artery calcification (CAC) score (Agatston Units) assessed by non-contrast cardiac CT scans from baseline to 24 months follow-up and will be analyzed as continuous variable in the entire population.

### Secondary outcomes

The secondary outcomes are as follows:

- Change in CAC score from baseline to 24 months in two prespecified subgroups (baseline CAC score
   <400 and ≥ 400) (numerical)</li>
- Change in CAC score from baseline to 12 months and from 12 to 24 months, both for the full cohort as well as for the two subgroups (numerical)
- Change in plaque volume (mm³), composition and plaque burden parameter (%) on per-patient level assessed by contrast cardiac CT scans of total plaque, noncalcified plaque, low-attenuation noncalcified plaque and calcified plaque from baseline to 24 months (numerical)
- Change in presence of normal, non-obstructive and obstructive (>50% in left main stem or >70% in left anterior descending, left circumflex and right coronary arteries in segments >2 mm) coronary artery stenosis by visual assessment in contrast CT scans from baseline to 24 months (numerical)
- Number of patients with myocardial infarction, coronary revascularization and all-cause death in the two groups during the follow-up period (dichotomous)

### Planned tables and figures and corresponding analyses

### Table 1. Characteristics of patients at baseline

Statistical methods applied for table 1 are similar to the statistics used for table 1 in the primary publication.

| Characteristics | Vitamin K +D | Placebo | p-value |
|-----------------|--------------|---------|---------|
| | group | group | |

| | (N=XX) | (N=XX) |
|--------------------------------------------------------|--------|--------|
| Age – years [numerical] | | |
| Body-mass index [numerical] | | |
| Coexisting condition – no (%) | | |
| Diabetes | | |
| Hyperlipidemia | | |
| Hypertension | | |
| Atrial fibrillation | | |
| Renal failure, eGFR < 60 mL/min1.73 m <sup>2</sup> | | |
| Family history of premature CVD | | |
| Smoking status | | |
| Active smokers - no (%) | | |
| Former smokers – no (%) | | |
| Non-smokers – no (%) | | |
| HDL – mmol/L | | |
| LDL – mmol/L | | |
| Total cholesterol – mmol/L | | |
| Estimated GFR – ml/min/1.73 m <sup>2</sup> [numerical] | | |
| dp-ucMGP – pmol/L | | |
| Systolic blood pressure – mmHg [numerical] | | |
| Diastolic blood pressure – mmHg [numerical] | | |
| Medications – no (%) | | |
| ACE inhibitor or ARB | | |
| Beta-blocker | | |
| Mineralocorticoid-receptor antagonist | | |
| Antiplatelet therapy | | |
| NOAC | | |
| Statin therapy | | |
| Baseline CAC score – AU [numerical] | | |
| Total population | | |
| < 400 AU | | |
| ≥ 400 AU | | |

ACE denotes angiotensin-converting enzyme, ARB angiotensin-receptor blocker, AVC aortic valve calcification, CAC coronary artery calcification, dp-ucMGP dephosphorylated-uncarboxylated Matrix Gla-Protein, GFR glomerular filtration rate, HDL high-density lipoprotein, LDL low-density lipoprotein, NOAC new-onset anticoagulant

<sup>†</sup> The body-mass index is the weight in kilograms divided by the square of the height in meters.

### Table 2. Primary outcome – main and secondary analyses

Statistical methods applied for table 2 are similar to the statistics used for table 2 in the primary publication. The main analysis is on mean change and treatment effect from baseline to 24 months follow-up. Secondary analyses as shown in the table are derived from the same statistical model.

| | Mean cha<br>from 0 to<br>months ( | 12 | Mean cha<br>from 12 t<br>months ( | o 24 | Mean cha<br>from 0 to<br>months ( | 24 | Treatment<br>effect<br>from 0 to<br>12<br>months<br>(95% CI) | Treatment<br>effect<br>from 12 to<br>24<br>months<br>(95% CI) | Treatment<br>effect<br>from 0 to<br>24<br>months<br>(95% CI) | p-value <sup>a</sup> | p-value <sup>b</sup> | p-value <sup>c</sup> | p-value <sup>d</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Vitamin | Placebo | Vitamin | Placebo | Vitamin | Placebo | | | | | | | |
| | K+D | group | K+D | group | K+D | group | | | | | | | |
| CAC score | group | | group | | group | | | | | | | | |
| (Continuou | | | | | | | | | | | | | |
| s AU) | | | | | | | | | | | | | |
| CAC score | | | | | | | | | | | | | |
| (baseline | | | | | | | | | | | | | |
| CAC score | | | | | | | | | | | | | |
| < 400 AU) | | | | | | | | | | | | | |
| CAC score | | | | | | | | | | | | | |
| (baseline | | | | | | | | | | | | | |
| CAC score | | | | | | | | | | | | | |
| ≥ 400 AU) | | | | | | | | | | | | | |

p-value<sup>a</sup> for the treatment effect from baseline to 12 months follow-up
p-value<sup>b</sup> for the treatment effect from 12 to 24 months follow-up
p-value<sup>c</sup> for the treatment effect from baseline to 24 months follow-up
p-value<sup>d</sup> for the difference in treatment effect from the first 12 months to last 24 months

### Table 3. Analyses on plaque composition and – burden in the total cohort

Analyses on change from baseline to 24 months on per patient level in all participants will be carried out similar to Table 2.

| | Vitamin K+D group | Placebo group | Group difference | |
|---|---|---|---|---|
| | Mean change from baseline (95 % CI) | Mean change<br>from baseline<br>(95 % CI) | Treatment effect<br>(95 % CI) | p-value |
| Plaque volume and | d composition | • | | |
| Total plaque (mm³) | | | | |
| Calcified plaque (mm³) | | | | |
| Noncalcified plaque (mm³) | | | | |
| Low-attenuation<br>noncalcified<br>plaque (<30 HU)<br>(mm³) | | | | |
| Plaque burden | | | | |
| Total plaque<br>burden (%) | | | | |
| Calcified plaque (%) | | | | |
| Noncalcified plaque (%) | | | | |
| Low-attenuation<br>noncalficied<br>plaque (<30 HU)<br>(%) | | | | |

### Table 4. Analysis on coronary obstruction

Change in frequency of level of coronary obstruction (no/nonobstructive/obstructive) from baseline to 24 months will be compared between treatment groups by mixed-effects ordered logistic regression including a random intercept for each patient and a fixed effects interaction between treatment and time point. As baseline measurements are obtained before randomization, treatment at baseline will be modelled as a separate common treatment category, constraining baseline measurements to no systematic treatment effect between the two treatment arms, as suggested in literature (6).

| Baseline | 24 months follow-up | Group difference |
|----------|---------------------|------------------|

| | Vitamin K+D<br>group | Placebo<br>group | Vitamin K+D<br>group | Placebo<br>group | Treatment effect OR | p-value |
|---|---|---|---|---|---|---|
| | | | | | (95% CI) | |
| Coronary obstruct | tion | | | | | |
| Normal – no (%) | | | | | | |
| Nonobstructive | | | | | | |
| – no (%) | | | | | | |
| Obstructive – no | | | | | | |
| (%) | | | | | | |
| Total | | | | | | |
| 1 vessel | | | | | | |
| 2 vessel | | | | | | |
| 3 vessel | | | | | | |

### Table 5. Analysis on cardiovascular events

Events from baseline to 24 months follow-up will be reported as counts and proportions and will be compared between groups by logistic regression estimating OR with 95% CI.

| | Vitamin K+D group | group Placebo group Group diffe | | erence |
|---|---|---|---|---|
| | Number (%) | Number (%) | OR (95% CI) | p-value |
| Events | | | | |
| Myocardial infarction | | | | |
| PCI procedure | | | | |
| CABG surgery | | | | |
| All cause death | | _ | | |

### Supplementary table S1. Adjusted analyses of the primary outcome

Results from an adjusted analysis of the primary outcome, mean change in CAC score from baseline to 24 months follow-up. The analysis will be performed as a regression adjusting for known cardiovascular risk factors (those included in Table S1) to further investigate the treatment effect.

| | Coefficient change baseline to 24 months (95% CI) | p-value |
|---|---|---|
| Intervention (Vitamin K+D) | | |
| Predictor variable | | |
| Age, yrs | | |
| BMI, kg/m <sup>2</sup> | | |
| Diabetes | | |
| Hyperlipidemia | | |
| Hypertension | | |
| Atrial fibrillation | | |
| Renal failure | | |
| Family history of premature CVD | | |
| Smoking status | | |

| Former smoker |
|--------------------|
| Active smoker |
| CAC score ≥ 400 AU |

### Supplementary table S2. Analysis on compliant patients

Analysis on patients with compliance > 90% from baseline to 24 months.

| | | Vitamin K +D group | Placebo group | Group difference | 2 |
|---|---|---|---|---|---|
| | | Number<br>(proportion) | Number<br>(proportion) | Odds ratio (95<br>% CI) | P-value |
| Compliance of at | t least 90% | (proportion) | (ргорогион) | NA NA | |
| | | Mean change from baseline (95 % CI) | Mean change<br>from baseline<br>(95 % CI) | Treatment<br>effect (95 % CI) | P-value |
| Primary outcome | Primary outcome (only including with compliance of at least 90%) | | | | |
| Continuous<br>CAC score | | | | | |

### Supplementary table S3. Stratified analyses of the primary outcome

Stratified analyses for mean change in CAC score for the total population from baseline to 24 months follow-up in this table are similar to the statistics used for table 5 in the primary publication.

| | Vitamin K+D group | Placebo group | | |
|---|---|---|---|---|
| | Mean change from baseline (95 % CI) | Mean change from baseline (95 % CI) | Treatment effect (95 % CI) | p-value |
| Age < 70 years | | | | |
| Age ≥70 years | | | | |
| No diabetes | | | | |
| Diabetes | | | | |
| No<br>hyperlipidemia<br>Hyperlipidemia<br>No hypertension | | | | |
| Hypertension | | | | |
| No atrial fibrillation | | | | |
| Atrial fibrillation | | | | |
| No renal failure | | | | |
| Renal failure | | | | |
| Non-smoker | | | | |

| Active/former |
|-------------------|
| smoker |
| No statin therapy |
| Statin therapy |
| dp-ucMGP (below |
| median) |
| dp-ucMGP (above |
| median) |

Supplementary table S4. Analyses on difference in the two groups at baseline, 12 and 24 months

| | Baseline 12 mon | | 12 month | S | 24 months | | p-<br>value <sup>a</sup> | p-<br>value <sup>b</sup> | p-<br>value <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|
| | Vitamin<br>K+D<br>group | Placebo<br>group | Vitamin<br>K+D<br>group | Placebo<br>group | Vitamin<br>K+D<br>group | Placebo<br>group | | | |
| Plaque volum | | position | <b>U</b> = - | <u> </u> | <b>U</b> | <u>I</u> | I. | <u>I</u> | |
| Total<br>plaque<br>(mm³) | | | | | | | | | |
| Calcified plaque (mm³) | | | | | | | | | |
| Noncalcified plaque (mm³) | | | | | | | | | |
| Low-<br>attenuation<br>noncalcified<br>plaque (<30<br>HU) (mm³) | | | | | | | | | |
| Plaque burde | n | • | | • | | • | • | • | • |
| Total<br>plaque<br>burden (%) | | | | | | | | | |
| Calcified plaque (%) | | | | | | | | | |
| Noncalcified plaque (%) | | | | | | | | | |
| Low-<br>attenuation<br>noncalcified<br>plaque (<30<br>HU) (%) | | | | | | | | | |

p-value<sup>a</sup> for the difference in change from baseline to 12 months follow-up

p-value  $^{\rm b}$  for the difference in change from 12 to 24 months follow-up

p-value<sup>c</sup> for the difference in change from baseline to 24 months follow-up

### Supplementary tables S5, S6. Analyses on plaque composition and – burden in the two subgroups

| Participants with CAC score < 400 | Vitamin K+D group | Placebo group | Group difference | |
|---|---|---|---|---|
| AU | Mean change from | Mean change | Treatment effect | P-value |
| | baseline (95 % CI) | from baseline<br>(95 % CI) | (95 % CI) | |
| Plaque volume and | d composition | | | • |
| Total plaque | | | | |
| (mm³) | | | | |
| Calcified plaque | | | | |
| (mm³) | | | | |
| Noncalcified | | | | |
| plaque (mm³) | | | | |
| Low-attenuation | | | | |
| noncalcified | | | | |
| plaque (<30 HU) | | | | |
| (mm³) | | | | |
| Plaque burden | | | | |
| Total plaque | | | | |
| burden (%) | | | | |
| Calcified plaque | | | | |
| (%) | | | | |
| Noncalcified | | | | |
| plaque (%) | | | | |
| Low-attenuation | | | | |
| noncalcified | | | | |
| plaque (<30 HU) | | | | |
| (%) | | | | |

| Participants with CAC score ≥ 400 | Vitamin K+D group | Placebo group | Group difference | |
|---|---|---|---|---|
| AU | Mean change from baseline (95 % CI) | Mean change<br>from baseline<br>(95 % CI) | Treatment effect<br>(95 % CI) | P-value |
| Plaque volume and | d composition | 1 (55 % 5.) | l | |
| Total plaque (mm³) | | | | |
| Calcified plaque (mm³) | | | | |
| Noncalcified plaque (mm³) | | | | |

| Low-attenuation |
|------------------|
| noncalcified |
| plaque (<30 HU) |
| (mm³) |
| Plaque burden |
| T |
| Total plaque |
| burden (%) |
| Calcified plaque |
| (%) |
| Noncalcified |
| plaque (%) |
| Low-attenuation |
| noncalcified |
| plaque (<30 HU) |
| (%) |

Figure 1. Enrolment and Randomization of Patients.

\* Excluded due to known CVD, including MI, PCI and CABG procedure



### Figure 2. CAC score progression according to treatment allocation.

CAC score at baseline, 12, and 24 months will be presented as line graph for the two treatment groups presenting mean with 95% confidence interval (as obtained from the linear mixed models applied for Table 3). Moreover it will be presented for the two subgroups (CAC score < 400 and ≥400 AU). (See mockup figure 2A below, 2B and 2C are similar)



Figure 3. Change in plaque volume from baseline to 24 months

Change in plaque volume (mm<sup>3</sup>) with the 4 groups (total, calcified, noncalcified, low-attenuation noncalcified plaque) from baseline to 24 months follow-up will be presented as a box plot to show difference between the treatment group and placebo group.



Figure 4. Forest plot of stratified analyses of the primary outcome

Coefficients with 95% confidence intervals from stratified analyses (as reported in Table 4) for differences in primary outcome (change of CAC score from baseline to 24 months) between treatment groups will be presented as a forest plot. (See mockup figure below.)



### Planned analyses for secondary publication: Changes in volumetric bone mineral density in the lumbar spine and total hip

#### Exclusion criteria

Participants with use of prednisolone, anti-osteoporotic drugs, and patients with metabolic bone diseases (such as: prostate cancer, bone metastatic cancers, myelotomies, rheumatoid arthritis, primary hyperparathyroidism), patient with immobilization during observation will be excluded.

### **Outcomes**

### Primary outcome

- Co-primary outcome 1: change in BMD in spine from baseline to 24 month (numerical)
- Co-primary outcome 1: change in BMD in hip from baseline to 24 month (numerical)

### Secondary outcomes

The secondary outcomes are as follows:

- Trabecular vBMD; total hip, femoral neck, inter- and subtrochanteric regions
- Cortical vBMD; total hip, femoral neck, inter- and subthrocanteric regions
- Cortical bone geometry and microstructure:
  - o Cortical area; total hip, femoral neck, inter- and subtrochanteric regions
  - Mean Cortical thickness femoral neck; femoral neck is evaluated in 16 sectors, and mean cortical thickness is calculated and the sum of all sectors divided by 16.
- Trabecular bone geometry
  - o Trabecular area; total hip, femoral neck, inter- and subtrochanteric regions
- Estimated bone strength:
  - o Hip Cross sectional Moment of Intertia (CSMI)
  - Hip Section Modulus

### Planned tables and figures and corresponding analyses

### Table 1. Characteristics of patients at baseline

Statistical methods applied for table 1 are similar to the statistics used for table 1 in the primary publication.

| Characteristics | Vitamin K +D | Placebo | p-value |
|---|---|---|---|
| | group | group | |
| | (N=XX) | (N=XX) | |
| Age – years [numerical] | | | |
| Body-mass index [numerical] | | | |
| Height [numerical] | | | |
| Weight [numerical] | | | |
| Coexisting condition – no (%) | | | |
| Diabetes | | | |
| Renal failure, eGFR < 60 mL/min1.73 m <sup>2</sup> | | | |
| Cancer | | | |
| Thyroid disease | | | |
| Fracture history (yes/no) – no (%) | | | |
| Calcium intake (mg) [numerical] | | | |
| Smoking status | | | |
| Active smokers - no (%) | | | |
| Former smokers – no (%) | | | |
| Non-smokers – no (%) | | | |
| Estimated GFR – ml/min/1.73 m² [numerical] | | | |
| dp-ucMGP – pmol/L | | | |
| Vitamin D | | | |
| Calcium | | | |
| Medications – no (%) | | | |
| Prednisolon | | | |
| Eltroxin | | | |
| Thycapzol | | | |

dp-ucMGP dephosphorylated-uncarboxylated Matrix Gla-Protein, GFR glomerular filtration rate, † The body-mass index is the weight in kilograms divided by the square of the height in meters.

### Table 2. Main analyses

Primary and secondary numerical outcomes will be analyzed by mixed effects linear regression. The mixed effects linear regression models will include a fixed effect for treatment, a fixed effect for time point (baseline and 24 months) and a fixed effects interaction between treatment and time point. As baseline measurements are obtained before randomization, treatment at baseline will be modelled as a separate common treatment category, constraining baseline measurements to no systematic treatment effect between the two treatment arms, as suggested in literature (6). All mixed effects models will include a random intercept for each included patient. Normality assumptions on residuals and random effects will be evaluated by normal quantile-quantile plots. In case deviations from normality assumptions are detected analyses will be repeated with nonparametric bootstrapping with 1,000 bootstrapping samples (handling individual patients as bootstrapping clusters, and treatment groups as bootstrapping strata).

Missing data will be excluded from analyses in Table 2 (but see sensitivity analyses below).

Table 2 might be split into multiple tables in the resulting manuscript to ease dissemination.

| | | Vitamin K +D | Placebo | | |
|---|---|---|---|---|---|
| | | group | | | |
| | | Mean change | group<br>Mean change | Treatment effect | P-value |
| | | (95 % CI) | Mean change<br>(95 % CI) | (95 % CI) | r-value |
| Primary outcomes | | (33 % CI) | (33 /0 CI) | (33 /0 CI) | 1 |
| Volumetric BMD in | 0 – 24 months | | | | |
| spine | 0 – 24 months | | | | |
| Volumetric BMD in | 0 – 24 months | | | | |
| hip | 0 – 24 months | | | | |
| Secondary outcomes | | | | | |
| Volumetric bone minera | I density (mg/cm3) | | | | |
| voidifietric borie miliera | ruensity (mg/cms) | | | | |
| Trabeculært vBMD | 0 – 24 months | | | | |
| total hip | | | | | |
| Trabeculært vBMD | 0 – 24 months | | | | |
| femoral neck | | | | | |
| Trabeculært vBMD | 0 – 24 months | | | | |
| inter-trochanteric | | | | | |
| regions | | | | | |
| Trabeculært vBMD | 0 – 24 months | | | | |
| sub-trochancheric | | | | | |
| regions | | | | | |
| Cortical vBMD total | 0 – 24 months | | | | |
| hip | | | | | |
| Cortical vBMD | 0 – 24 months | | | | |
| femoral neck | | | | | |
| Cortical vBMD inter- | 0 – 24 months | | | | |
| trochanteric regions | | | | | |
| Cortical vBMD sub- | 0 – 24 months | | | | |
| trochancheric | | | | | |
| regions | | | | | |
| Bone geometry (cm2) | | 1 | | | 1 |
| Trabecular area sub- | 0 – 24 months | | | | |
| trochancheric | | | | | |
| regions | | | | | |
| Trabecular area | 0 – 24 months | | | | |
| femoral neck | | | | | |
| Trabecular area | 0 – 24 months | | | | |
| inter-trochanteric | | | | | |
| regions | | | | | |
| Trabecular area sub- | 0 – 24 months | | | | |
| trochancheric | | | | | |
| regions | | | | | |
| Cortical area sub- | 0 – 24 months | | | | |
| trochancheric | | | | | |
| regions | | | | | |
| Cortical area | 0 – 24 months | | | | |
| femoral neck | | | | | |

| Cortical area inter-<br>trochanteric regions | 0 – 24 months |
|----------------------------------------------|---------------|
| Cortical area sub- | 0 – 24 months |
| trochancheric | |
| regions | |
| Bone microstructure ( | cm) |
| Cortical thickness | 0 – 24 months |
| sub-trochancheric | |
| regions | |
| Cortical thickness | 0 – 24 months |
| femoral neck | |
| Cortical thickness | 0 – 24 months |
| inter-trochanteric | |
| regions | |
| Cortical thickness | 0 – 24 months |
| sub-trochancheric | |
| regions | |
| Estimated bone strength | |
| CSMi (cm4) | 0 – 24 months |
| Section Modulus | 0 – 24 months |
| (cm3) | |

### Supplementary Table S1. Sensitivity analysis: Primary outcome with imputation

If more than 5% of observations are missing at 24 months for the main analysis of the primary outcomes reported in Table 2 the analysis will be repeated using multiple imputation (assuming missing at random) by linear regression with all baseline characteristics included in Table 1 as covariates generating 100 imputation sets. Results will be reported in a table structured as Table 2.

### Supplementary Table S2. Main analyses adjusted for baseline characteristics

Main analysis as included in Table 2 will be repeated adjusted for D vitamin level and calcium intake at baseline as numerical covariates. The adjusted results will reported in a table structured as Table 2.

### Supplementary Table S3. Mean and standard deviation of outcomes at baseline and 24 months

Mean and standard deviation (SD) for all outcomes stratified by treatment group will be reported at baseline and at 24 months.

| | Baseline | | 24 months | |
|---|---|---|---|---|
| | Vitamin K +D Placebo group | | Vitamin K +D | Placebo group |
| | group | | group | |
| | Mean (SD) | Mean (SD) | Mean (SD) | Mean (SD) |
| Primary outcomes | | | | |
| Volumetric BMD in | | | | |
| spine | | | | |

| Volumetric BMD in | | |
|----------------------|-----------------------|----|
| hip | | |
| Secondary outcome | S | |
| Volumetric bone mi | neral density (mg/cm3 | 3) |
| Trabeculært vBMD | | |
| total hip | | |
| Trabeculært vBMD | | |
| femoral neck | | |
| Trabeculært vBMD | | |
| inter-trochanteric | | |
| regions | | |
| Trabeculært vBMD | | |
| sub-trochancheric | | |
| regions | | |
| Cortical vBMD | | |
| total hip | | |
| Cortical vBMD | | |
| femoral neck | | |
| Cortical vBMD | | |
| inter-trochanteric | | |
| regions | | |
| Cortical vBMD | | |
| sub-trochancheric | | |
| regions | | |
| Bone geometry (cm2 | 2) | |
| Trabecular area | | |
| sub-trochancheric | | |
| regions | | |
| Trabecular area | | |
| femoral neck | | |
| Trabecular area | | |
| inter-trochanteric | | |
| regions | | |
| Trabecular area | | |
| sub-trochancheric | | |
| regions | | |
| Cortical area sub- | | |
| trochancheric | | |
| regions | | |
| Cortical area | | |
| femoral neck | | |
| Cortical area inter- | | |
| trochanteric | | |
| regions | | |
| Cortical area sub- | | |
| trochancheric | | |
| regions | (cm) | |
| Bone microstructure | e (Cifi) | |

| Cortical thickness |
|-------------------------|
| sub-trochancheric |
| regions |
| Cortical thickness |
| femoral neck |
| Cortical thickness |
| inter-trochanteric |
| regions |
| Cortical thickness |
| sub-trochancheric |
| regions |
| Estimated bone strength |
| CSMi (cm4) |
| Section Modulus |
| (cm3) |

Figure 1. Enrollment and Randomization of Patients.

Flow chart



### Figure 2. Change in BMD (spine and hip) from baseline to 24 months

Change in BMD spine and BMD hip from baseline to 24 months follow-up will be presented as a box plots to show difference between the treatment group and placebo group.



Figure 3. Calcium intake from baseline to 24 months

Calcium intake from baseline to 24 months follow-up will be presented as line graph for the two treatment groups presenting mean with 95% confidence interval obtained by fitting a linear mixed model specified as those applied for numerical outcomes in the main publication. Calcium intake is calculated as:

200 + (number of units milk x 200)+(number of units chees x 200)+(number of units fermented milk x 200)



### References

- 1. Lindholt JS, Frandsen NE, Fredgart MH, Øvrehus KA, Dahl JS, Møller JE, et al. Effects of menaquinone-7 supplementation in patients with aortic valve calcification: study protocol for a randomised controlled trial. BMJ Open. 2018;8(8):e022019.
- 2. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)—A metadata-driven methodology and workflow process for providing translational research informatics support. Journal of Biomedical Informatics. 2009;42(2):377-81.
- 3. Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, et al. The REDCap consortium: Building an international community of software platform partners. Journal of Biomedical Informatics. 2019;95:103208.
- 4. Stata Statistical Software: Release 16. 16 ed. College Station, TX: StataCorp LLC; 2019.
- 5. Levene H. Robust tests for equality of variances. Robust Tests for Equality of Variances. 1960:278-92.
- 6. J T, L B, T H, J R, M W, M H. Different ways to estimate treatment effects in randomised controlled trials. Contemp Clin Trials Commun. 2018;10:80-5.